CLINICAL TRIAL: NCT07115069
Title: Conduct of the REsponses in Function and Outcomes From RYGB vs. Medication Study (REFORM) Study by Research Coordinators
Brief Title: Comparison of Body Composition Changes With Weight Loss Interventions
Acronym: REFORM
Status: Recruiting | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Jason Samuels, Principal Investigator, Vanderbilt University Medical Center
Other Study IDs: 251035; U16066 (Other: Vanderbilt University Medical Center)
Record Dates: First submitted 2025-07-25; First posted 2025-08-11 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-08

CONDITIONS: Obesity
Keywords: obesity; GLP-1 receptor agonist; gastric bypass surgery; bariatric surgery; incretin; glucagon like peptide 1 receptor agonist; robotic surgery
MeSH Terms: conditions — Obesity | interventions — semaglutide; Tirzepatide; Laparoscopy; Robotics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- GLP-1 Receptor Agonists Arm: Patient recieving Glucagon Like Peptide 1 Receptor Agonists (GLP1RA) or incretin polyagonists.
  Interventions: Drug: GLP-1 receptor agonist
- Gastric Bypass surgery (laparoscopic): Patients undergoing gastric bypass laparoscopically
  Interventions: Procedure: Gastric Bypass Surgery (laparoscopic)
- Gastric Bypass surgery (robotic): Patients undergoing Gastric Bypass surgery robotically
  Interventions: Procedure: Gastric Bypass Surgery (robotic)

INTERVENTIONS:
Drug: GLP-1 receptor agonist — Any FDA-approved GLP-1 receptor agonist
  Other Names: semaglutide; tirzepatide
  Groups: GLP-1 Receptor Agonists Arm
Procedure: Gastric Bypass Surgery (laparoscopic) — Patients undergo laparoscopic gastric bypass with a roux limb between 75 - 150 cm and biliopancreatic limb between 50 - 150 cm as determined by the primary surgeon.
  Other Names: RNYGB
  Groups: Gastric Bypass surgery (laparoscopic)
Procedure: Gastric Bypass Surgery (robotic) — Patients undergo robotic gastric bypass with a roux limb between 75 - 150 cm and biliopancreatic limb between 50 - 150 cm as determined by the primary surgeon.
  Other Names: RNYGB
  Groups: Gastric Bypass surgery (robotic)

SUMMARY:
This study is being done to compare the effects of a newer class of weight loss medications to weight loss surgery on the body's muscle, metabolism, and side effects over time. People with severe obesity often lose weight using either medications like GLP-1 receptor agonists (such as semaglutide or tirzepatide) or by having bariatric surgery, such as gastric bypass. While both approaches can lead to weight loss, they may affect the body in different ways.

The investigators are inviting adult patients who are planning to either start one of these weight loss medications or undergo gastric bypass surgery to join this study. Participants will be asked to complete four body composition scans (called DXA scans) over the course of a year-at the beginning of the study and again at 3, 6, and 12 months. These scans will help us measure changes in fat and muscle. Participants will also complete surveys and provide information on side effects, such as nausea or fatigue, that may affect their eating or activity levels.

The investigators' goal is to better understand how different weight loss treatments impact not just weight, but also muscle mass, energy levels, and side effects. This information may help doctors and patients choose the most appropriate treatment in the future.

DETAILED DESCRIPTION:
Patients are benefiting from landmark advancements in obesity treatments with the advent of Glucagon-like Peptide 1 Receptor agonists (GLP1RA) such as semaglutide and tirzepatide, which achieve weight loss of 15-20% in clinical trials.2,4,21 However, numerous questions surround the safety and efficacy of GLP1RAs compared to established surgical interventions. Minimally Invasive gastric bypass (GB) remains the benchmark for obesity treatments, with superior weight loss of 25-35%, and an extensive body of literature demonstrating long-term safety and efficacy, with rare complications and dramatic improvements in obesity-related comorbidities and quality of life.22,23 To date, an absence of guidelines exists to guide patients and clinicians in appropriate selection of therapies for obesity, largely resulting from the lack of head-to-head comparison for safety and efficacy of these interventions.

GLP1RAs carry several risks potentially limiting their benefit. The appetite suppression induced by GLP1RAs may result in disproportionate skeletal muscle depletion, the magnitude of which remains incompletely characterized.24,25 Loss of skeletal muscle can lead to poorer functional outcomes despite weight loss, and may lead to sarcopenic obesity if weight regain occurs after drug cessation.7,10 Additionally, a majority of patients taking GLP1RAs report adverse gastrointestinal (GI) symptoms including nausea, vomiting, constipation and abdominal pain, with reported discontinuation rates of >50% in clinical practice.26-29 Furthermore, the significant cost of GLP1RAs (averaging $10,000-15,000 annually) has placed considerable strain on healthcare systems. Recent studies suggest long-term cost benefits of GB over GLP1RAs30, but more research is needed to further delineate the most effective strategy in terms of both clinical outcomes and economic impact.

This study aims to compare impact of GLP1RAs and GB on skeletal muscle composition, GI symptom profiles, and quality of life metrics. This study will also compare changes in GI symptoms and quality of life between patients undergoing laparoscopic versus robotic GB.

Specific Aim 1: Compare change in appendicular lean body mass (LBM) after GLP-1 receptor agonists & gastric bypass at 3, 6, and 12 months. Utilizing Dual-Energy X-ray Absorptiometry (DXA) scans conducted prior to surgery or mediation initiation and 3-, 6-, and 12-months post-intervention, the investigators will quantify the ratio of LBM loss to total weight loss with GLP1RAs and GB surgery. The investigators hypothesize that GLP1RA treatment will result in greater proportional loss of LBM than GB after 12 months of treatment. Data will be analyzed using mixed-effects models accounting for baseline characteristics and intervention type.

Specific Aim 2: Compare GI symptoms changes and overall quality of life following gastric bypass vs GLP1RAs and investigate real-world tolerability of GLP1RAs. Utilizing the validated Patient Assessment of Upper Gastrointestinal Disorders Symptoms Questionnaire (PAGI-SYM), administered at baseline and monthly intervals for 6 months, this study will compare the trajectory and severity of GI symptoms between those receiving GLP1RA and those who undergo GB. The investigators hypothesize that GLP1RA treatment will result in higher (worse) PAGI-SYM scores than GB throughout the study period. Additionally, will measure Health Related Quality of Life (HRQOL) monthly from intervention to 6 months post-intervention and compare trajectory of overall HRQOL after GLP1RA and GB.

Specific Aim 3: Comparison of GI symptoms and quality of life changes at 3 and 6 mo with robotic surgery and GLP1RA therapies. The investigators will also study how robotic GB compares to GLP1RA therapy in terms of GI symptomatology and health-related quality of life (HRQOL). HRQOL will be assessed using the validated SF-36 and the obesity-specific IWQOL-Lite instruments at baseline, 3 months, 6 months, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥35 and ≤60
* Primary weight loss surgery (gastric bypass), or
* Medical weight loss with GLP1RAs (Semaglutide or Tirzepatide)

Exclusion Criteria:

* Revisional gastric bypass (e.g. sleeve to bypass),
* <3 months of continuous use of GLP1RA,
* Type 1 Diabetes,
* Myocardial Infarction,
* Unstable Angina or Heart Failure,
* Stroke
* Solid organ transplantation,
* Systemic glucocorticoid prior 28 days,
* Uncontrolled Hypertension, (Systolic > 150, Diastolic > 90)
* Untreated Hyperthyroidism
* Chronic Kidney Disease (EGFR < 60).

Ages: 21 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants seeking medical or surgical weight loss for class III obesity
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-08-09 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Skeletal Muscle Loss | 6 months
  loss of skeletal muscle (reported as appendicular lean body mass (LBM) on DXA) as a percent total body mass loss from baseline to 6 months as determined by DXA
Skeletal Muscle Loss | 12 months
  loss of skeletal muscle (reported as appendicular lean body mass (LBM) on DXA) as a percent total body mass loss from baseline to 12 months as determined by DXA
Patient Assessment of Upper Gastrointestinal Disorders Symptoms Questionnaire | 6 months
  Median Patient Assessment of Upper Gastrointestinal Disorders Symptoms Questionnaire (PAGI-SYM score). Scores are on a 6 point Likert scale 0 (none/absent) to 5 (very severe) symptoms.
Patient Assessment of Upper Gastrointestinal Disorders Symptoms Questionnaire | 12 months
  Median Patient Assessment of Upper Gastrointestinal Disorders Symptoms Questionnaire (PAGI-SYM score). Scores are on a 6 point Likert scale 0 (none/absent) to 5 (very severe) symptoms.

SECONDARY OUTCOMES:
Incidence of 10% weight loss | 6 months
  Number of patients achieving ≥10% total body weight loss
Incidence of 10% weight loss | 12 months
  Number of patients achieving ≥10% total body weight loss
Incidence of 15% weight loss | 6 months
  Number of patients achieving ≥15% total body weight loss
Incidence of 15% weight loss | 12 months
  Number of patients achieving ≥15% total body weight loss
Grip Strength | 3, 6, and 12 months
  Change in Grip strength measured by Jamar Grip Strength Hydraulic Dynanometer.
PAGI-SYM sub-scale scores | 6 months
  Sub-scale scores: 1. heartburn/regurgitation, 2. nausea/vomiting, 3. postprandial fullness, 4. bloating, 5. upper and lower abdominal pain

CONTACTS AND LOCATIONS:
Overall Officials: Jason M Samuels, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Any sharing of de-identified data for scientific dissemination (e.g., publications, presentations) will comply with federal guidance and institutional requirements.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: At least 5 years after study end